CLINICAL TRIAL: NCT04684472
Title: Phase I, Open Label, Study of CXCR4 Modified CD19 CAR-T Therapy in Patients With Relapsed or Refractory CD19+ B-cell Malignancies
Brief Title: Modified CD19 CAR-T in Patients With Relapsed or Refractory CD19+ B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liqun Zou (Other)
Responsible Party: Sponsor-Investigator, Liqun Zou, Professor of Department of Medical Oncology, Sichuan University
Organization: Sichuan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCART-003
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Leukemia
Keywords: Modified CD19 CAR-T
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified anti-CD19 CAR T cell therapy (Experimental): CAR T cell therapy
  Interventions: Biological: Modified anti-CD19 CAR T cells

INTERVENTIONS:
Biological: Modified anti-CD19 CAR T cells — intravenous infusion

SUMMARY:
This study aims to evaluate the safety and tolerance of modified CD19 CAR T cells in treating refractory/relapsed B-cell malignancies. CAR-T cells will be investigated as a single agent both in relapsed/refractory B-cell acute lymphoblastic leukaemia (B-ALL) and up to 60% of patients with B-cell non-Hodgkin's lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-70 years;
2. Estimated survival time ≥ 12 weeks;
3. Histologically confirmed diagnosis of CD19+ B-ALL or CD19+ B-NHL(meeting one of the following conditions):

   1. Ineffectively or relapses after 2 or more remedial treatments
   2. Relapse after auto-HSCT or unsuitable for auto-HSCT;
4. At least one assessable tumor lesion;
5. ECOG performance status 0 to 2;
6. Creatinine clearance rate≥ 60 ml/min, ALT and AST ≤ 2.5 times of upper limit of normal, total bilirubin ≤ 1.5 times of upper limit of normal;
7. Male and female of reproductive potential must agree to use birth control during the study and for at least 30 days post study;
8. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients with other uncontrolled malignancies;
2. Previously treated with any CAR-T cell product or other genetically-modified T cell therapy;
3. Patients with HIV infection, hepatitis B (HBsAg positive) or hepatitis C（anti-HCV positive);
4. Patients with central nervous system involvement by lymphoma ,malignant cells in cerebrospinal fluid or history of brain metastasis;
5. Patients with atrial or ventricular involvement by B-cell malignancies;
6. Patients with tumor mass require urgent treatment, such as ileus or vascular compression;
7. Patients with severe disease or other uncontrolled diseases that were not suitable for this trial, such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, grade 2-3 hypertension;
8. Unstable pulmonary embolism, deep venous embolism, or other major arterial/venous thromboembolism events occurred within 30 days prior to randomization. If patients receive anticoagulant therapy, the treatment dose must be stable prior to randomization;
9. Any situations that the investigators believes were not suitable for this trial;
10. Long-term use of immunosuppressive agents after organ transplantation, except for the patients recently or currently receiving inhaled steroids;
11. Pregnant(or lactation) women;
12. Patients with severe active infections(excluding simple urinary tract infection and bacterial pharyngitis)within 30 days prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [Safety and Tolerability] | Up to 5 years after modified CD19 CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Dose-limiting toxicity (DLT) | Baseline up to 28 days after modified CD19 CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
B-cell malignancies, Overall response rate(ORR) | 3 months, 6 months
  Assessment of ORR(ORR=CR+PR)
B-cell malignancies, Overall survival | Up to 2 years after modified CD19 CAR-T cells infusion
  From the first infusion of modified CD19 CAR-T cells to death or the last visit
B-cell malignancies, progression-free survival（PFS） | Up to 2 years after modified CD19 CAR-T cells infusion
  From the first infusion of modified CD19 CAR-T cells to the occurrence of any event, including death, relapse, disease progression, and the last visit
B-cell malignancies, disease control rate (DCR) | Month 6,12,18 and 24
  Assessment of DCR(DCR=CR+PR+SD)

CONTACTS AND LOCATIONS:
Overall Officials: liqun zou, phd, Principal Investigator — Sichuan University
Locations (1):
- Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No